CLINICAL TRIAL: NCT04483791
Title: A Non-Randomized, Clinical Registry of the Dynamx Novolimus Eluting Coronary Bioadaptor System in the Treatment of Patients With De Novo Native Coronary Artery Lesions
Brief Title: DynamX Bioadaptor Hong Kong Registry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ELX-CL-2001
Record Dates: First submitted 2020-07-16; First posted 2020-07-23 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting stent; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — novolimus

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, multicenter registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DynamX Novolimus Eluting Coronary Bioadaptor System (Other): DynamX use in de novo coronary artery lesions
  Interventions: Combination Product: DynamX Novolimus Eluting Coronary Bioadaptor System

INTERVENTIONS:
Combination Product: DynamX Novolimus Eluting Coronary Bioadaptor System — up to two de novo native coronary artery lesions measuring between 2.25 and 3.5 mm in diameter and<=34 mm in length receiving the DynamX Novolimus Eluting Coronary Bioadaptor System
  Other Names: Novolimus; Bioadaptor

SUMMARY:
Prospective, non-randomized, multicenter registry

DETAILED DESCRIPTION:
Enrollment of up to 50 subjects with up to two de novo native coronary artery lesions measuring between 2.25 and 3.5 mm in diameter and<=34 mm in length receiving the DynamX Novolimus Eluting Coronary Bioadaptor System (CSS), with primary, interim clinical follow-up via telephone at 1 month. Follow-up will continue at 6, and 12 months. to capture cardiovascular related hospitalizations related to the study devic

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18 and ≤ 80 years
2. Subject (or legal guardian) understands the trial requirements and treatment procedures and provides written informed consent prior to any trial-specific tests or treatment
3. Indication for a percutaneous intervention with stent implantation in native epicardial arteries including patients with stable coronary artery disease and acute coronary syndromes (non-ST-elevated myocardial infarction)
4. Vessel diameter (2.25-3.5 mm) and lesions length ≤ 34 mm suitable for implantation using a single stent per lesion
5. All lesions requiring PCI should be amendable for implantation with the study stent
6. Successful pre-dilatation of the first lesion defined as no waist in the inflated pre-dilatation balloon using two orthogonal views using a pre- dilatation balloon diameter size ranging from the reference vessel diameter to 0.25 mm smaller than the reference vessel diameter, and a residual diameter stenosis prior to study device implantation by visual estimate being < 35%

Exclusion Criteria:

1. Target lesion / vessel specific

   1. Lesions in the left main
   2. Venous or arterial bypass grafts
   3. In-stent restenosis
   4. Chronic total occlusion
   5. Ostial lesions (< 3 mm from the ostium of the RCA, LAD or Cx)
   6. Stent implanted < 10 mm from the target lesion in the previous 30 days.
   7. Lesion requiring rotablation or atherectomy because of, but not limited to severe calcification
   8. Bifurcation lesions requiring a planned 2 or more stent technique
2. Patient specific:

   1. STEMI
   2. Acute myocardial infarction with Killip Class III and IV
   3. Known LVEF < 30%
   4. Life expectancy < 1 year
   5. Patients on renal dialysis or known GFR < 30 ml/min
3. Planned surgery necessitating interruption of dual antiplatelet therapy within the first 6 months
4. Known intolerance to components of the investigational product or medication required (e.g. intolerance to concomitant anticoagulation or antiplatelet therapy)
5. Subject is receiving or will require chronic anticoagulation therapy (e.g. coumadin, dabigatran, apixaban, rivaroxaban, edoxaban or low molecular weight heparin)
6. Subject is currently participating in another clinical trial with an investigational drug or device that has not yet completed its primary endpoint
7. Known pregnancy or breastfeeding
8. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Kwong Wah Hospital, Hong Kong, Kowloon
  - Queen Elizabeth Hospital, Hong Kong, Kowloon
  - Queen Mary Hospital, Hong Kong, Pok Fu Lam
  - Chinese University of Hong Kong / Prince of Wales Hospital, Hong Kong, Sha Tin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of up to 50 subjects with up to two de novo native coronary artery lesions measuring between 2.25 and 3.5 mm in diameter and ≤ 34 mm in length receiving the DynamX Novolimus Eluting Coronary Bioadaptor System (CBS), with primary, interim clinical follow-up via telephone at 1 month. Follow-up will continue at 6, and 12 months. to capture cardiovascular related hospitalizations related to the study device.
Period: Overall Study
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Started | 50
Completed | 49
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 50
Diabetes Mellitus [Count of Participants; unit: Participants] | 18
Hypertension [Count of Participants; unit: Participants] | 39
Hypercholesterolemia/Dyslipidemia [Count of Participants; unit: Participants] | 46
Smoking (previous or current) [Count of Participants; unit: Participants] | 29
Prior myocardial infarction (MI) [Count of Participants; unit: Participants] | 6
Prior percutaneous coronary intervention [Count of Participants; unit: Participants] | 9
Stable angina [Count of Participants; unit: Participants] | 20
Unstable angina [Count of Participants; unit: Participants] | 20
ST Elevation MI [Count of Participants; unit: Participants] | 2
Non-ST Elevation MI [Count of Participants; unit: Participants] | 4
Silent ischemia / Asymptomatic [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Acute Device Success
Description: Percentage of patients with an attainment of a final result of < 30% residual stenosis using the DynamX bioadaptor with standard pre-dilatation and post-dilatation (if applicable) catheters
Time Frame: Immediately after final stent placement (intraprocedure)
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 49

2. Primary Outcome: Device Oriented Clinical Endpoint; Number of Participants With Cardiovascular Death, Target Vessel Myocardial Infarction (TV-MI) or Clinically-Driven Target Lesion Revascularization (CD-TLR).
Description: the composite of cardiovascular death, target vessel myocardial infarction or clinically-driven target lesion revascularization
Time Frame: 12 Months
Population: 49 out of 50 participants enrolled were evaluated at the 12-month visit related to 1 lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 49
Participants | 0

3. Secondary Outcome: Device Oriented Clinical Endpoint; Number of Participants With Cardiovascular Death, Target Vessel Myocardial Infarction (TV-MI) or Clinically-Driven Target Lesion Revascularization (CD-TLR).
Description: as for outcome 2
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Number of Participants With Cardiovascular and Non-Cardiovascular Death
Description: cardiac and non-cardiac
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

5. Secondary Outcome: Number of Participants With Cardiovascular and Non-Cardiovascular Death
Description: cardiac and non-cardiac
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

6. Secondary Outcome: Number of Participants With Cardiovascular and Non-Cardiovascular Death
Description: cardiac and non-cardiac
Time Frame: 12 months
Population: 49 out of 50 participants enrolled were evaluated at the 12-month visit related to 1 lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 49
Participants | 0

7. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: target vessel and non-target vessel
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

8. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: target vessel and non-target vessel
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

9. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: target vessel and non-target vessel
Time Frame: 12 months
Population: 49 out of 50 participants enrolled were evaluated at the 12-month visit related to 1 lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 49
Participants | 0

10. Secondary Outcome: Number of Participants With Clinically-Indicated Target Lesion Revascularization
Description: clinically-indicated
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

11. Secondary Outcome: Number of Participants With Clinically-Indicated Target Lesion Revascularization
Description: clinically-indicated
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

12. Secondary Outcome: Number of Participants With Clinically-Indicated Target Lesion Revascularization
Description: clinically-indicated
Time Frame: 12 month
Population: 49 out of 50 participants enrolled were evaluated at the 12-month visit related to 1 lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 49
Participants | 0

13. Secondary Outcome: Device Oriented Clinical Endpoint; Number of Participants With Cardiovascular Death, Target Vessel Myocardial Infarction (TV-MI) or Clinically-Driven Target Lesion Revascularization (CD-TLR).
Description: as for outcome 2
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
Number analyzed (Participants) | 50
Participants | 0

ADVERSE EVENTS:
Time Frame: Through 12-months
Arm/Group | DynamX Novolimus Eluting Coronary Bioadaptor System
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 30/50
Other Adverse Events (participants affected / at risk) | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DynamX Novolimus Eluting Coronary Bioadaptor System (N=50)
Procedure Complications (Injury, poisoning and procedural complications) | 3
Arrhythmia requiring treatment (Cardiac disorders) | 5
Recurrent ischemia/chest pain (Cardiac disorders) | 5
Hypertension (Cardiac disorders) | 2
Hypotension/Syncope (Cardiac disorders) | 2
Chest Infection (Infections and infestations) | 1
Bleeding Complications/Hematoma (General disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7
Extremity Pain/Injury (General disorders) | 2
Renal/UT Events (Renal and urinary disorders) | 1
Heart Failure (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DynamX Novolimus Eluting Coronary Bioadaptor System (N=50)
Arrhythmia requiring treatment (Cardiac disorders) | 1
Recurrent Ischemia/Chest Pain (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 1
Bleeding complications/hematoma (General disorders) | 1
Other non-cardiac events (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04483791/Prot_001.pdf